CLINICAL TRIAL: NCT00396032
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Tenecteplase for Restoration of Function in Dysfunctional Hemodialysis Catheters
Brief Title: A Study of Tenecteplase for Restoration of Function in Dysfunctional Hemodialysis Catheters
Acronym: TROPICS 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N3700g
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-06-03 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-05

CONDITIONS: Dysfunctional Hemodialysis Catheters
Keywords: HD; Hemodialysis; Catheter clearance; TNKase; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tenecteplase
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — For the initial treatment, 2 mL of placebo instilled into each lumen of the HD catheter; subsequent treatments were 2 mL of open-label tenecteplase
  Arms: 2
Drug: tenecteplase — For the initial treatment, 2 mL of reconstituted lyophilized tenecteplase instilled into each lumen of the HD catheter; subsequent treatments were 2 mL of open-label tenecteplase
  Arms: 1

SUMMARY:
This was a Phase III, randomized, double-blind, placebo-controlled study conducted at 37 centers in the United States. 150 subjects ≥ 16 years of age who required hemodialysis (HD) and had a dysfunctional HD catheter were enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable, in the opinion of the investigator
* Use of a cuffed, tunneled HD catheter
* HD prescribed at a BFR of ≥300 mL/min
* Baseline BFR (at any time during the first 60 minutes of HD) of <300 mL/min at an associated pre-pump negative arterial pressure in the range between and including -240 mmHg and -280 mmHg
* Baseline BFR (at any time during the first 60 minutes of HD) at least 25 mL/min below the prescribed BFR
* Demonstrated BFR of ≥300 mL/min (using catheter lines in the customary direction) at an arterial pressure in the range of 0 to -280 mmHg in at least one HD session in the 14 days prior to Visit 1
* Anticipated use of the same catheter for at least four consecutive HD sessions, on the same type and model of HD apparatus
* Able to have fluids infused at the volume necessary to instill study drug into the HD catheter

Exclusion Criteria:

* HD catheter with sustainable BFR of ≥300 mL/min following subject repositioning
* HD catheter inserted <2 days prior to screening
* Evidence of a mechanical, non-thrombotic cause of HD catheter dysfunction (e.g., kink in the catheter or suture constricting the catheter) or dysfunction caused by known fibrin sheath
* Use of an implantable port
* HD catheter that is internally coated with any therapeutic agent (e.g., the Decathlon™ Gold catheter)
* Anticipated use of catheter for any other type of diagnostic or therapeutic procedure (i.e., other than HD) during study drug treatment
* Previously treated in this study or any tenecteplase catheter clearance trial
* Use of any investigational drug or therapy (defined as any drug or therapy that is not FDA approved) within 28 days prior to screening
* Use of a fibrinolytic agent (e.g., alteplase, tenecteplase, reteplase, or urokinase) within 7 days prior to Visit 1
* Known to be pregnant or breastfeeding at screening or at Visit 1
* Known bacteremia or known or suspected infection in the HD catheter
* Known history of any of the following: intracranial hemorrhage (within the previous 3 years), intracranial aneurysm, or arteriovenous malformation
* Use of heparin (unfractionated or low molecular weight) or other anticoagulants (e.g., for the treatment of heparin-induced thrombocytopenia) within 24 hours prior to Visit 1, except for heparin used only during HD or for prophylaxis (e.g., heparin lock or deep vein thrombosis prophylaxis)
* Subjects treated with warfarin only: international normalized ratio (INR) >3.0 within 7 days prior to Visit 1, or a target INR range that allows for an INR >3.0 A laboratory test to confirm the INR must have been performed within 7 days prior to Visit 1.
* Initiation of or increase in dose of Plavix® (clopidogrel bisulfate) within 7 days prior to Visit 1
* Hemoglobin ≥12.0 g/dL if on an erythropoiesis-stimulating agent (e.g., darbepoetin or erythropoietin) and the dose of the erythropoiesis-stimulating agent has not been held or reduced per institutional policy
* At high risk for bleeding events or embolic complications (i.e., recent pulmonary embolus, deep vein thrombosis, endarterectomy, or clinically significant right-to-left shunt) in the opinion of the investigator, or with known condition for which bleeding constitutes a significant hazard
* BFR of <300 mL/min because of symptomatic hypotension
* Uncontrolled hypertension in the opinion of the investigator
* Known hypersensitivity to tenecteplase or any component of the formulation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gillespie, M.D., FASN, Study Director

REFERENCES:
- [Derived] Tumlin J, Goldman J, Spiegel DM, Roer D, Ntoso KA, Blaney M, Jacobs J, Gillespie BS, Begelman SM. A phase III, randomized, double-blind, placebo-controlled study of tenecteplase for improvement of hemodialysis catheter function: TROPICS 3. Clin J Am Soc Nephrol. 2010 Apr;5(4):631-6. doi: 10.2215/CJN.06520909. Epub 2010 Feb 4. PMID 20133491

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was randomized but not treated, therefore the modified intent-to-treat (MITT) analysis population was 149.
Groups:
- Tenecteplase: For the initial treatment, 2 mL of reconsituted lyophilized tenecteplase instilled into each lumen of the HD catheter; subsequent treatments were 2 mL of open-label tenecteplase
Period: Overall Study
Arm/Group | Tenecteplase | Placebo
Started | 74 | 76
Completed | 70 | 71
Not Completed | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase | Placebo | Total
Number analyzed (Participants) | 74 | 75 | 149
Age, Customized [Number; unit: participants]
  < 17 years | 0 | 0 | 0
  >= 17 years to < 65 years | 44 | 51 | 95
  >= 65 years | 30 | 24 | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.1) | 57.8 (16.5) | 59.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Had Treatment Success With Respect to Blood Flow Rate (BFR) at Visit 1
Description: Treatment success is defined as BFR of ≥300 mL/min and an increase from baseline BFR of ≥25 mL/min at an associated target arterial pressure in the range of 0 to -280 mmHg 30 (±10) minutes prior to the end of HD and at the end of HD.
Time Frame: Visit 1 of HD treatment
Population: Modified intent to treat (MITT) population
Measure: Number; unit: percentage of success
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 74 | 75
percentage of success | 21.6 | 5.3
Statistical Analysis 1: Comparison: Tenecteplase vs Placebo; Test type: Superiority or Other; p = 0.0044, Cochran-Mantel-Haenszel — Stratified by baseline BFR: 0-199 mL/min, 200-274 mL/min, and 275-299 mL/min
Statistical Analysis 2: Comparison: Tenecteplase vs Placebo; Test type: Superiority or Other; p = 0.0035, Chi-squared

2. Primary Outcome: Incidence of Targeted Adverse Events (AEs) From Initial Study Drug Administration Through the Start of Visit 2
Description: Targeted AEs were intracranial hemorrhages (ICHs), major bleeding, embolic events, thrombosis, catheter-related bloodstream infections (CRBSIs), and catheter related complications
Time Frame: Visits 1 and 2 of consecutive HD treatments
Population: MITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 74 | 75
percentage of participants
  Intracranial hemorrhage | 0 | 0
  Major bleeding | 0 | 0
  Embolic event | 0 | 0
  Thrombosis | 0 | 0
  Catheter-related blood stream infection | 0 | 4.0
  Catheter-related complication | 0 | 0

3. Secondary Outcome: Change in BFR From Baseline to the End of HD at Visit 1
Description: BFR is measured in mL/minute.
Time Frame: Visit 1 of HD treatment
Population: MITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 74 | 75
percentage of participants
  < 0 mL/min | 8.1 (102.97) | 9.3 (55.98)
  0-24 mL/min | 58.1 | 80.0
  25-49 mL/min | 8.1 | 2.7
  50-99 mL/min | 8.1 | 4.0
  100-149 mL/min | 5.4 | 1.3
Statistical Analysis 1: Comparison: Tenecteplase vs Placebo; Test type: Superiority or Other; p = 0.0396, Cochran-Mantel-Haenszel — Stratified by baseline BFR: 0-199 mL/min, 200-274 mL/min, and 275-299 mL/min

4. Secondary Outcome: Percentage of Subjects Who Had Treatment Success With Respect to BFR at Visit 2 (MITT Population With Extended Dwell Tenecteplase at Visit 1)
Description: as for outcome 1
Time Frame: Visit 2 of consecutive HD treatments
Population: MITT population with extended-dwell tenecteplase at Visit 1
Measure: Number; unit: percentage of success
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 24 | 39
percentage of success | 41.7 | 38.5

5. Secondary Outcome: Percentage of Subjects Who Had Treatment Success With Respect to BFR at Visit 2 (MITT Population With Open-label Tenecteplase at Visit 2)
Description: as for outcome 1
Time Frame: Visit 2 of consecutive HD treatments
Population: MITT population with open-label tenecteplase at Visit 2
Measure: Number; unit: percentage of success
Arm/Group | Tenecteplase | Placebo
Number analyzed (Participants) | 26 | 23
percentage of success | 11.5 | 34.8

ADVERSE EVENTS:
Time Frame: The AEs/SAEs were recorded through the completion of Visit 4.
Description: Safety-evaluable population.
  SAEs of hypoclycemia and convulsion occurred in the placebo group after treatment with open-label tenecteplase.
  Note: The incidence of each AE/SAE is reported as the number of participants experiencing the event, not the number of occurrences for each AE/SAE.
Arm/Group | Tenecteplase | Placebo
Serious Adverse Events (participants affected / at risk) | 1/74 | 5/75
Other Adverse Events (participants affected / at risk) | 12/74 | 11/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=74) | Placebo (N=75)
Bacteraemia (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (N=74) | Placebo (N=75)
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Stomach Discomfort (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Catheter Related Complication (General disorders) | 1 | 0
Catheter Site Pain (General disorders) | 1 | 0
Catheter Site Pruritus (General disorders) | 1 | 0
Catheter Thrombosis (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Feeling Cold (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Thrombosis in Device (Injury, poisoning and procedural complications) | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Renal and urinary disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.